CLINICAL TRIAL: NCT01424800
Title: Influence of Variations in Systemic Blood Flow and Blood Pressure on Cerebral Oxygenation Measured by Cerebral Oximetry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2011/208
Record Dates: First submitted 2011-08-22; First posted 2011-08-29 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Cerebral Oxygen Saturation
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- change in blood pressure and blood flow (Experimental): 34 patients will form the experimental group, in which changes of blood pressure and blood flow will be induced and monitored.
  Interventions: Device: A disposable NIRS (near-infrared spectroscopy) sensor will be applied on the patient's forehead for continuous registration of the cerebral oxygen saturation.

INTERVENTIONS:
Device: A disposable NIRS (near-infrared spectroscopy) sensor will be applied on the patient's forehead for continuous registration of the cerebral oxygen saturation. — When the patient is on CPB, pressure and/or flow will be changed while continuously measuring ScO2. Temperature, CO2 , arterial oxygen content, hematocrit and anesthesia will be kept constant during the measurements. First, baseline MAP (mean arterial pressure), baseline ScO2 and baseline central venous oxygen saturation (SvO2) are determined. With the interventions, we will induce a change of 20% in MAP and/or flow. This is within the normal range during operations. Changes in blood pressure will be obtained by the use of vasoactive agents (sodiumnitroprusside for blood pressure decrease and phenylephrine for blood pressure increase). Flow is regulated by manual control of the pump flow. Values of the different variables will be obtained after a 5 min stabilisation period. Flow/pressure interventions will be randomized.

SUMMARY:
This study emphasizes on the influence of changes in systemic flow and systemic mean arterial blood pressure (MAP) during cardiopulmonary bypass (CPB) on cerebral oxygenation assessed by near-infrared spectroscopy (NIRS). The aim of the study is to determine whether variations in systemic flow, in MAP, or in both variables at the same time have the greatest impact on the cerebral oxygen saturation.

DETAILED DESCRIPTION:
Cerebral autoregulation is defined as the whole of regulatory mechanisms that maintains a constant cerebral blood flow (CBF) during changes in cerebral perfusion pressure (CPP). Cerebrovascular resistance adjusts when CPP changes in order to keep CBF constant. In contrast with this concept of pressure-mediated autoregulation, it is suggested that cerebral autoregulation is focused on maintaining homeostasis of the cerebral metabolic rate of oxygen (CMRO2). We assume that both flow and pressure contribute to the regulation of CMRO2.

Assessment of cerebral oxygenation - Cerebral oxygen saturation will be monitored with near-infrared spectroscopy (NIRS). NIRS allows simple, continuous and non-invasive measurement of cerebral oxygen saturation (ScO2)and primarily cerebral venous saturation. Cerebral oxygen saturation will be monitored with a FDA-approved devices: INVOS 5100 (Somanetics Corporation, Troy, MI, USA).

To study the effects of changes in pressure and in flow, we need a condition where we can alter these variables separately and in a controlled manner. Therefore this study will be performed during cardiopulmonary bypass (CPB). Pressure will be varied with the administration of routinely used vasoactive substances, while flow will be varied by altering the pump flow manually. We hypothesize that if we change one parameter (pressure or flow), a compensatory mechanism will preserve the CMRO2 homeostasis, with no change in ScO2. On the other hand, if we change both pressure and flow, we expect a significant effect on cerebral oxygen saturation. With 20 % changes in pressure and/or flow, we expect a change in NIRS values of approximately 5 %. Previous studies showed that this kind of reduction is well tolerated by the brain. This means that the proposed changes are within the normal physiological range, and will have no adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-100 years, scheduled for elective cardiac surgery, written informed consent.

Exclusion Criteria:

* History of cerebrovascular disease or symptomatic carotid artery stenosis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Blood flow | during the entire surgery
  Changes in blood flow during cerebral oxygen saturation measured with NIRS, during surgery when the patient is on cardiopulmonary bypass.
Blood pressure | during the entire surgery
  Changes in blood pressure during cerebral oxygen saturation measured with NIRS, during surgery when the patient is on cardiopulmonary bypass.

CONTACTS AND LOCATIONS:
Overall Officials: Annelies Moerman, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium